CLINICAL TRIAL: NCT02240732
Title: Surgical Tourniquets and Cerebral Emboli Pilot Study
Brief Title: Surgical Tourniquets and Cerebral Emboli
Status: Completed | Type: Observational
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Principal Investigator, Victoria Gibbs, Doctor, University Hospitals Coventry and Warwickshire NHS Trust
Other Study IDs: STCE2.0
Record Dates: First submitted 2014-09-15; First posted 2014-09-16 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis; RA; Trauma
MeSH Terms: conditions — Osteoarthritis; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Total knee replacement patients: Patients who are due to have a total knee replacement will be studied to look for the presence of Emboli.
  Observational with imaging.

SUMMARY:
BACKGROUND In 2012 76,497 primary total knee (TKR) replacements were performed in England, Wales and Northern Ireland . Traditionally TKR surgery is undertaken with the aid of a surgical tourniquet. A surgical tourniquet is an occlusive device applied around a patient's leg. The tourniquet squeezes the leg (including blood vessels within the leg) and can therefore reduce the amount of bleeding that occurs while it is inflated. An intraoperative tourniquet can therefore help to improve the surgical field of view. Although the majority of surgeons prefer to undertake TKR surgery using a tourniquet a small but increasing number are now not pursuing these devices.

There is robust evidence that the risk of deep vein thrombosis is increased if a tourniquet is used for TKR surgery. In addition embolic material in the venous system have been observed following TKR surgery and have been noted to be present in the right atrium with transoesophageal (TOE) echo intra-operatively. , Significant and potentially life threatening emboli have been documented to enter the cerebral circulation via pulmonary arterio-venous shunts and patent foramen ovale (PFO) (27% of patients at autopsy) , . The clinical manifestations of cerebral emboli post tourniquet deflation in TKR are not fully understood. Fat embolism syndrome and post-operative confusion in TKR patients may be the result of emboli formed during a TKR. ,

AIM

* Is there evidence of emboli entering the cerebral circulation following tourniquet deflation in TKR surgery?
* Is there evidence of MRI detectable brain lesions and or any clinical change in cognition compared in patients undergoing TKR surgery with a tourniquet compared to those that do not have a tourniquet?

ELIGIBILITY:
Inclusion Criteria:

* i.Aged >18
* ii.Undergoing elective TKR
* iii.Able to give written informed consent
* iv.No contraindications to MR imaging

Exclusion Criteria:

* i. Ages <16
* ii. Not able to give written informed consent
* iv. Contraindications to MR imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are due to have a total knee replacement.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of Emboli on Transcranial Doppler | Intra-operative
  2 independent technicians will verify the number of emboli detected. Non-invasive
MRI brain scan - presence of Emboli | Post-operatively, prior to discharge
  Reviewed by Professor of radiology - presence, number and volume of diffusion weighted lesions

SECONDARY OUTCOMES:
Mini-mental state examination | Pre-operative vs Post-operative
  Set of 30 questions which test cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Gibbs, BA, MBBS, Principal Investigator — UHCW
Locations (1):
- University Hospital Warwickshire and Coventry, Coventry, United Kingdom

REFERENCES:
- [Background] Tai TW, Lin CJ, Jou IM, Chang CW, Lai KA, Yang CY. Tourniquet use in total knee arthroplasty: a meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2011 Jul;19(7):1121-30. doi: 10.1007/s00167-010-1342-7. Epub 2010 Dec 15. PMID 21161177
- [Background] Parmet JL, Horrow JC, Pharo G, Collins L, Berman AT, Rosenberg H. The incidence of venous emboli during extramedullary guided total knee arthroplasty. Anesth Analg. 1995 Oct;81(4):757-62. doi: 10.1097/00000539-199510000-00017. PMID 7574006
- [Background] Parmet JL, Berman AT, Horrow JC, Harding S, Rosenberg H. Thromboembolism coincident with tourniquet deflation during total knee arthroplasty. Lancet. 1993 Apr 24;341(8852):1057-8. doi: 10.1016/0140-6736(93)92414-o. PMID 8096961
- [Background] Arroyo JS, Garvin KL, McGuire MH. Fatal marrow embolization following a porous-coated bipolar hip endoprosthesis. J Arthroplasty. 1994 Aug;9(4):449-52. doi: 10.1016/0883-5403(94)90057-4. PMID 7964778
- [Background] Pugsley W, Klinger L, Paschalis C, Treasure T, Harrison M, Newman S. The impact of microemboli during cardiopulmonary bypass on neuropsychological functioning. Stroke. 1994 Jul;25(7):1393-9. doi: 10.1161/01.str.25.7.1393. PMID 8023354
- [Background] Riding G, Daly K, Hutchinson S, Rao S, Lovell M, McCollum C. Paradoxical cerebral embolisation. An explanation for fat embolism syndrome. J Bone Joint Surg Br. 2004 Jan;86(1):95-8. PMID 14765873
- [Background] Caillouette JT, Anzel SH. Fat embolism syndrome following the intramedullary alignment guide in total knee arthroplasty. Clin Orthop Relat Res. 1990 Feb;(251):198-9. PMID 2295174